CLINICAL TRIAL: NCT06854692
Title: In-game Cervical Exercises to Reduce Subsequent Post-game Decrease of Shoulder Internal Rotation Range of Motion and External Rotation Strength in Baseball Pitchers
Brief Title: Impact of Cervical Exercises During Simulated Game on Throwing Shoulder Motion and Strength
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sacred Heart University (Other)
Responsible Party: Principal Investigator, Jason Grimes, PT, PhD, OCS, ATC, Associate Professor, Sacred Heart University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IRB-FY2025-188
Record Dates: First submitted 2025-02-20; First posted 2025-03-03 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Shoulder
Keywords: shoulder; throwing athlete; range of motion; strength; cervical retraction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental)
  Interventions: Other: Cervical retraction exercise
- Control group (No Intervention)

INTERVENTIONS:
Other: Cervical retraction exercise — Participants will perform end-range cervical retraction and cervical retraction with extension, holding the end-range of motion for 3 seconds and performing 10 repetitions of each exercise.
  Arms: Intervention group

SUMMARY:
The goal of this clinical trial is to investigate the impact of performing cervical exercises during a simulated game on shoulder range of motion and strength in collegiate baseball picthers. The main questions it aims to answer are:

Can performing cervical retraction/extension exercises help to maintain shoulder internal rotation range of motion in the throwing shoulder after a pitching session? Can performing cervical retraction/extension exercises help to maintain shoulder external rotation strength in the throwing shoulder after a pitching session?

Researchers will compare the effects of cervical retraction/extension exercises to no exercise to see if shoulder range of motion or strength is impacted.

Participants will perform end-range cervical retraction and cervical retraction with extension, holding the end-range of motion for 3 seconds and performing 10 repetitions of each exercise between each inning of a simulated 5-inning game.

DETAILED DESCRIPTION:
Glenohumeral internal rotation deficit (GIRD) and rotator cuff weakness have been identified as predisposing factors in sustaining a shoulder or elbow injury in pitchers. The appearance of GIRD in symptomatic throwers has been attributed to osseous adaptations as well as soft tissue restrictions of the posterior capsule, deltoid and posterior cuff. Trakis identified that those adolescent pitchers with pain complaints had presented with weakness of the posterior shoulder musculature. Tyler noted preseason supraspinatus weakness was significantly associated with an increase in shoulder and elbow injury risk in high school pitchers. Despite studies indicating a correlation with rotator cuff weakness and injury, there is a lack of consensus on the underlying cause of the rotator cuff weakness.

The presentation of GIRD and rotator cuff weakness typically occurs in tandem and a question arises if these are linked, and if they might actually occur in response to the act of throwing. A subsequent loss of internal rotation range of motion and weakness of external rotation has been noted immediately following pitching. In a study of 67 asymptomatic professional pitchers, Reinold found a significant loss of passive shoulder internal rotation (IR) immediately following pitching that was also evident 24 hours after throwing. Reinold purported that the altered range of motion may be related to acute musculotendinous adaptations in response to the eccentric muscle activity of the external rotators during the throwing motion. Gandhi found a decrease in external rotation strength and a statistically and clinically significant decrease in voluntary muscle activation of the infraspinatus immediately following pitching in a simulated game. His contention was that the weakness was due to incomplete neuromuscular recruitment.

The posterior rotator cuff demonstrates large electromyographic (EMG) activity during the act of throwing. Overused muscle shortens over time, changing the muscle length-tension properties and becoming more readily active and weaker after time. The cause of the weakness may be neuro-reflexive or structural in nature. The combination of loss of IR and weakness of the external rotators might be explained by the concept of "tightness weakness" as described by Janda. The author's propose that the loss of shoulder internal rotation range of motion and external rotation strength may be linked and centrally mediated from the cervical spine. The act of throwing will produce a compressive force in the mid-cervical spine related to the compensatory movement of cervical extension, lateral flexion and rotation towards the throwing side. Pheasant demonstrated a decrease in shoulder external rotator strength following a maintained postural position of forward head and rounded shoulders for only 5 minutes. He noted that the resultant lower cervical flexion that accompanies the forward head posture can create foraminal stenosis at C4-C5, thereby causing a compression of the C5 nerve root.

In a case series, Pheasant demonstrated an increase in external rotation strength and resolution of pain complaints in 2 overhead athletes presenting with shoulder impingement by performing cervical retraction and cervical retraction with extension. He surmised that intermittent compression of the C5 nerve root could impair nerve function and ultimately cause rotator cuff weakness by affecting the suprascapular and axillary nerve that innervate the supraspinatus, teres minor and infraspinatus, and that the cervical retraction exercises reduced the compression. Internal rotation range of motion pre-intervention was only visually estimated and there was no indication of that motion being compared to the non-involved shoulder or if there was an improvement in motion following implementation of the exercises.

ELIGIBILITY:
Inclusion Criteria:

* an overhead thrower over the age of 18 years old
* currently painfree while throwing at their usual intensity

Exclusion Criteria:

* previous shoulder or elbow surgery on the throwing arm within the last 12 months
* currently in the post-operative phase of a shoulder or elbow surgery on the throwing arm
* currently participating in a rehabilitation program for shoulder or elbow pain
* currently not able to throw due to shoulder or elbow pain

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2025-05-31 (Actual); Primary Completion 2025-12-29 (Actual); Study Completion 2025-12-29 (Actual)

PRIMARY OUTCOMES:
Shoulder Internal Rotation ROM | Day 1
  measure of shoulder range of motion
Shoulder External Rotation Strength | Day 1
  measure of shoulder strength

CONTACTS AND LOCATIONS:
Locations (1):
- Sacred Heart University, Fairfield, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Paige P, Frank CC, Larnder R. (2010) Assessment and treatment of muscle imbalance: The Janda approach. Human Kinetics.
- [Background] Devaney LL, Denegar CR, Thigpen CA, Lepley AS, Edgar C, DiStefano LJ. Preseason Neck Mobility Is Associated With Throwing-Related Shoulder and Elbow Injuries, Pain, and Disability in College Baseball Pitchers. Orthop J Sports Med. 2020 May 18;8(5):2325967120920556. doi: 10.1177/2325967120920556. eCollection 2020 May. PMID 32523967
- [Background] Pheasant S, Haydt R, Gottstein T, Grasso A, Lombard N, Stone B. SHOULDER EXTERNAL ROTATOR STRENGTH IN RESPONSE TO VARIOUS SITTING POSTURES: A CONTROLLED LABORATORY STUDY. Int J Sports Phys Ther. 2018 Feb;13(1):50-57. PMID 29484241
- [Background] Pheasant S. CERVICAL CONTRIBUTION TO FUNCTIONAL SHOULDER IMPINGEMENT: TWO CASE REPORTS. Int J Sports Phys Ther. 2016 Dec;11(6):980-991. PMID 27904800
- [Background] Jobe FW, Tibone JE, Perry J, Moynes D. An EMG analysis of the shoulder in throwing and pitching. A preliminary report. Am J Sports Med. 1983 Jan-Feb;11(1):3-5. doi: 10.1177/036354658301100102. PMID 6829838
- [Background] Gandhi J, ElAttrache NS, Kaufman KR, Hurd WJ. Voluntary activation deficits of the infraspinatus present as a consequence of pitching-induced fatigue. J Shoulder Elbow Surg. 2012 May;21(5):625-30. doi: 10.1016/j.jse.2011.04.012. Epub 2011 Aug 10. PMID 21831667
- [Background] Reinold MM, Wilk KE, Macrina LC, Sheheane C, Dun S, Fleisig GS, Crenshaw K, Andrews JR. Changes in shoulder and elbow passive range of motion after pitching in professional baseball players. Am J Sports Med. 2008 Mar;36(3):523-7. doi: 10.1177/0363546507308935. Epub 2007 Nov 8. PMID 17991783
- [Background] Tyler TF, Mullaney MJ, Mirabella MR, Nicholas SJ, McHugh MP. Risk Factors for Shoulder and Elbow Injuries in High School Baseball Pitchers: The Role of Preseason Strength and Range of Motion. Am J Sports Med. 2014 Aug;42(8):1993-9. doi: 10.1177/0363546514535070. Epub 2014 Jun 3. PMID 24893778
- [Background] McClure P, Balaicuis J, Heiland D, Broersma ME, Thorndike CK, Wood A. A randomized controlled comparison of stretching procedures for posterior shoulder tightness. J Orthop Sports Phys Ther. 2007 Mar;37(3):108-14. doi: 10.2519/jospt.2007.2337. PMID 17416125
- [Background] Burkhart SS, Morgan CD, Kibler WB. The disabled throwing shoulder: spectrum of pathology Part I: pathoanatomy and biomechanics. Arthroscopy. 2003 Apr;19(4):404-20. doi: 10.1053/jars.2003.50128. PMID 12671624
- [Background] Crockett HC, Gross LB, Wilk KE, Schwartz ML, Reed J, O'Mara J, Reilly MT, Dugas JR, Meister K, Lyman S, Andrews JR. Osseous adaptation and range of motion at the glenohumeral joint in professional baseball pitchers. Am J Sports Med. 2002 Jan-Feb;30(1):20-6. doi: 10.1177/03635465020300011701. PMID 11798991
- [Background] Trakis JE, McHugh MP, Caracciolo PA, Busciacco L, Mullaney M, Nicholas SJ. Muscle strength and range of motion in adolescent pitchers with throwing-related pain: implications for injury prevention. Am J Sports Med. 2008 Nov;36(11):2173-8. doi: 10.1177/0363546508319049. Epub 2008 Jul 2. PMID 18596197
- [Background] Wilk KE, Macrina LC, Fleisig GS, Porterfield R, Simpson CD 2nd, Harker P, Paparesta N, Andrews JR. Correlation of glenohumeral internal rotation deficit and total rotational motion to shoulder injuries in professional baseball pitchers. Am J Sports Med. 2011 Feb;39(2):329-35. doi: 10.1177/0363546510384223. Epub 2010 Dec 4. PMID 21131681
- [Background] Garrison JC, Cole MA, Conway JE, Macko MJ, Thigpen C, Shanley E. Shoulder range of motion deficits in baseball players with an ulnar collateral ligament tear. Am J Sports Med. 2012 Nov;40(11):2597-603. doi: 10.1177/0363546512459175. Epub 2012 Sep 26. PMID 23019251